CLINICAL TRIAL: NCT02787642
Title: A Phase Ib Study of Olaparib With Concomitant Radiotherapy in Locally Advanced/Unresectable Soft-tissue Sarcoma
Brief Title: A Study of Olaparib With Concomitant Radiotherapy in Locally Advanced/Unresectable Soft-tissue Sarcoma
Acronym: RADIOSARP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB 2015-05; 2015-003722-13 (EudraCT Number)
Record Dates: First submitted 2016-05-02; First posted 2016-06-01 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Soft-tissue Sarcoma
Keywords: Advanced soft-tissue sarcoma; Unresectable Soft-tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olaparib in association with concomitant radiotherapy (Experimental): Olaparib will be administered per os bi-daily, as appropriate assigned dose level, during 7.5 weeks (D1 to D52). Olaparib should be started one week before the start of radiotherapy and will be continued until the last day of radiotherapy. Beyond this period, Olaparib could be continued at the investigator's discretion and after sponsor authorization, until progression. Radiotherapy consists of fractionated focal irradiation at a dose of 1.8 Grays (Gy) per fraction given once daily five days per week (Monday through Friday) over a period of 6.5 weeks, for a total dose of 59.4 Gy. Radiotherapy starts at D8.
  Interventions: Drug: Olaparib; Radiation: Concomitant Radiotherapy

INTERVENTIONS:
Drug: Olaparib — Olaparib will be administered per os bidaily, as appropriate assigned dose level, during 7.5 weeks (D1 to D52). Olaparib should be started one week before the start of radiotherapy and will be continued until the last day of radiotherapy. Beyond this period, Olaparib could be continued at the investigator's discretion and after sponsor authorization, until progression.
Radiation: Concomitant Radiotherapy — Radiotherapy consists of fractionated focal irradiation at a dose of 1.8 Grays (Gy) per fraction given once daily five days per week (Monday through Friday) over a period of 6.5 weeks, for a total dose of 59.4 Gy. Radiotherapy starts at D8.

SUMMARY:
A phase Ib study of Olaparib with concomitant radiotherapy in locally advanced/unresectable soft-tissue sarcoma.

DETAILED DESCRIPTION:
This is a multicenter, prospective phase Ib trial based on a dose escalation study design (3+3 traditional design) assessing four dose levels of Olaparib given with concomitant radiotherapy, followed by an expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Histology: patients with soft-tissue sarcoma histologically confirmed by central review (Pr Coindre team), except if the diagnosis was already confirmed by the RRePS Network,
2. Upper/Lower limb or trunk wall soft-tissue sarcoma,
3. Age ≥ 18 years,
4. Locally advanced or locally recurrent primitive tumor, outside any previously irradiated field. Patients presenting operable locally Advanced or lacally recurrent tumor can be included. Patients with metastases can be included.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2,
6. Life expectancy ≥ 6 months,
7. At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements,
8. Adequate hematological, renal, metabolic and hepatic function:

   * Haemoglobin ≥ 9 g/dL and no blood transfusions in the 14 days prior to study entry
   * Absolute neutrophil count (ANc) ≥ 1.5 x 109/L
   * Platelets ≥ 100 x 109/L
   * Total bilirubin ≤ 1.5 x upper limit of normality (ULN),
   * Alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) ≤ 2.5 x ULN,
   * Serum creatinine ≤ 150 μmol/L or creatinine clearance ≥ 50 mL/min (according to local institution) in case of serum creatinine > 150 μmol/L,
   * TP, INR ≤ 1.5 x ULN
9. Women of childbearing potential must have a negative serum pregnancy test within 28 days of study treatment, confirmed prior to treatment on day 1. Female patients of child bearing potential and their partners, who are sexually active, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for at least 1 month after last dose of study drug. Males patients, who are sexually active, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for at least 3 month after last dose of study drug. Acceptable birth control methods are described in appendix 10.

   Subjects of non-childbearing potential are those who have:
   * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments,
   * LH and FSH levels in the post menopausal range for women under 50,
   * radiation-induced oophorectomy with last menses >1 year ago,
   * chemotherapy-induced menopause with >1 year interval since last menses,
   * or surgical sterilisation (bilateral oophorectomy or hysterectomy).
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up,
11. Voluntary signed and dated written informed consent prior to any specific procedure,
12. Patients with a social security in compliance with the Law.

Exclusion Criteria:

1. Any previous treatment with a PARP inhibitor, including Olaparib,
2. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication,
3. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV) and are receiving antiviral therapy,
4. Patients with known active hepatic disease (i.e., Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids,
5. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, unstable spinal cord compression (untreated and unstable for at least 28 days prior to study entry), superior vena cava syndrome, extensive bilateral lung disease on HRCT scan or any psychiatric disorder that prohibits obtaining informed consent,
6. Patients with uncontrolled seizures,
7. Men or women of childbearing potential who are not using an effective method of contraception as previously describes; women who are pregnant or breast feeding,
8. No prior or concurrent malignant disease diagnosed or treated in the last 2 years, except for adequately treated in situ carcinoma of the cervix, basal or squamous skin cell carcinoma, or in situ transitional bladder cell carcinoma,
9. Patients receiving any systemic chemotherapy within 2 weeks from the last dose prior to study treatment (or a longer period depending on the defined characteristics of the agents used),
10. Concomitant use of known CYP3A4 inhibitors such as ketokonazole, itraconazole, ritonavir, indinavir, saquinavir, telithromycin, clarithromycin and nelfinavir,
11. Resting ECG with QTc > 470msec on 2 or more time points within a 24 hour period or family history of long QT syndrome,
12. Blood transfusions within 14 days prior to study start,
13. Patients with myelodysplastic syndrome/acute myeloid leukaemia,
14. Major surgery within 14 days of starting study treatment and patients must have recovered from any effects of any major surgery,
15. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
16. Patient unable to follow and comply with the study procedures because of any geographical, familial, social or psychological reasons,
17. Previous enrollment in the present study,
18. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
19. Patients who not have recovered from any effects of any major surgery
20. Individuals deprived of liberty or placed Under legal guardianship
21. Patients who have tumor in contact with, invading or encasing for more than 50% any major blood vessels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Olaparib evaluated up to six weeks after end of radiotherapy | Until to six weeks after end of radiotherapy

SECONDARY OUTCOMES:
Non-progression defined as CR, PR as per RECIST 1.1 | 6-month
Objective defined as CR or PR as per RECIST 1.1 | 6-month
Best objective response under treatment as per RECIST v 1.1 | End of treatment,an average of 6 months
Best response under treatment as per RECIST 1.1 | End of treatment,an average of 6 months
Progression-free survival (PFS) as per RECIST 1.1 | 1 year
Overall Survival (OS) | 1 year
Functional assessment graded using the Muskuloskeletal Tumour Society Rating Scale (Enneking, 1987) | Day 1, Week 8
Pharmacokinetics PK measurements expressed as the AUC of Olaparib | Weeks 1, 2, 5
Pharmacokinetics PK measurements expressed as half-life of Olaparib | Weeks 1, 2, 5
Pharmacokinetics PK measurements expressed as the concentration peak of Olaparib | Weeks 1, 2, 5

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Claudius Regaud - IUCT, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353